CLINICAL TRIAL: NCT01983397
Title: Effects of Two Physical Exercise Protocols on Cognition and Physical Performances in Oldest Old: a Randomized Controlled Trial
Brief Title: Effects of Two Physical Exercise Protocols on Cognition and Physical Performances in Elderly Over 80 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Juliana Hotta Ansai, Principal investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Ansai-01
Record Dates: First submitted 2013-10-31; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Sedentary
Keywords: aged, 80 and over; Exercise; Cognition; Balance; Randomized controlled trial
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resistance training (Experimental): Resistance training
  Interventions: Other: Resistance training
- Multicomponent training (Experimental): Multicomponent training
  Interventions: Other: Multicomponent training
- Control Group (No Intervention): The Control Group did not realize any intervention.

INTERVENTIONS:
Other: Multicomponent training — The multicomponent training consisted of individuals subjected to a multicomponent exercise program: 5 minute warm up, 20 minutes of aerobic exercise, 15-20 minutes of strength exercises, 10 minutes of coordination, agility and balance exercises and 5 minute of cool-down.
  Arms: Multicomponent training
Other: Resistance training — The resistance training was subjected to a strength training using weight machines adapted for elderly. The protocol followed three sets of 10 to 12 maximal repetitions, moderate speed (two seconds for the shortening phase and three seconds for the elongation phase) and one minute for rest interval between sets.
  Arms: Resistance training

SUMMARY:
The purpose of this study is to compare the effects of different trainings on cognition and physical performances in elderly over 80 years.

DETAILED DESCRIPTION:
Purpose: To compare the effects of 16-week multicomponent and resistance trainings on cognition and physical performances related to falls in oldest old people living in community; to analyze the same variables after 6-week detraining. Method: We conducted a randomized controlled trial with 69 community elderly over 80 years, sedentary and without cognitive disorder. Participants were allocated to control, multicomponent training or resistance training group. The multicomponent group performed a protocol involving warm-up, aerobic, strength, balance and cool-down exercises. The resistance group underwent to strength exercises using six machines: leg press, chest press, calf, back extension, abdominal and rowing. The control group did not perform any intervention. The trainings had progressive intensity, lasted 16 weeks and included three 1-hour sessions per week. The participants were evaluated at baseline, at the end of 16-week training and at 6-week detraining. The assessment consisted of anamnesis, depression (Geriatric Depression Scale), cognition (Montreal cognitive assessment), dual task walking (associated to cognitive and motor tasks), balance (unipedal and tandem tests), strength of lower limbs (sit-to-stand test) and history of falls. For statistical analysis by intention to treat, we adopted a significance level of α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* age between 80 and 95 years old
* live in community
* sedentary lifestyle
* ability to walk without help from another person with/without aid walking

Exclusion Criteria:

* any cardiovascular or infectious comorbidity described in the absolute contraindications of the Physical Activity Readiness Medical Examination
* Relative contraindications of cognitive, neurological and/or musculoskeletal comorbidities which make participation in protocols impossible
* Score in mini-state examination mental below the cutoff score designated by education level.

Ages: 80 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in lower limbs strength after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, after 16 weeks of training and 6 weeks of detraining
  Lower limbs strength was assessed by 5 times sit-to-stand test.
Changes from baseline in balance after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, after 16 weeks of training and 6 weeks of detraining
  Balance was assessed by unipedal test and tandem test.
Changes from baseline in dual task walking after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, after 16 weeks of training and 6 weeks of detraining
  Dual task was assessed by Timed Up and Go test with a cognitive task (speak day of week in reverse order) and motor task (carry a cup of water).
Changes from baseline in cognition after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, after 16 weeks of training and 6 weeks of detraining.
  Cognition was evaluated by Montreal Cognitive Assessment.

SECONDARY OUTCOMES:
Changes from baseline in number of falls after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, during 16 weeks of training and 6 weeks of detraining.
  Presence of falls was assessed by falls calendar and phone calls.
Changes from baseline in depression after 16 weeks of training and 6 weeks of detraining | Assessed at baseline, during 16 weeks of training and 6 weeks of detraining.
  Depression was assessed by abbreviated Geriatric Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana H Ansai, specialist, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil